CLINICAL TRIAL: NCT05332158
Title: The Adherence to Oral Anticoagulants and Statins Project
Brief Title: Medicines Gaps Study
Acronym: MeGa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Leeds Clinical Commissioning Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PH21/145969
Record Dates: First submitted 2022-01-18; First posted 2022-04-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Adherence, Medication; Statin Adverse Reaction; Anticoagulant Adverse Reaction
Keywords: adherence; barriers; anticoagulants; statins
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Masking Description: Researcher will be blinded to participants with pseudonymised data being collected for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): A single arm to administer questionnaires for patients barriers to adherence.
  Interventions: Behavioral: Questionnaires to report barriers to medication adherence

INTERVENTIONS:
Behavioral: Questionnaires to report barriers to medication adherence — One questionnaire specific to DOACs and one specific to statins have been integrated within the medical records system and will be sent to eligible patients to respond to following written informed consent.

SUMMARY:
The adherence project aims to understand adherence rates and barriers to Direct oral anticoagulants (DOACs) and statins and improve awareness of healthcare professionals on adherence across Leeds.

During the first component of the project, the investigation of rates of non-adherence was classed as service evaluation. The second component of this project, which this IRAS application refers to, will look into patient perspectives and barriers to adherence. Currently, such information is not routinely collected and only requested as part of shorter or longer consultations depending on a pre-defined clinical agenda and with little attention to adherence. Two specific questionnaires have been designed and integrated within the primary care medical records systems. Following invitation for target patients on DOACs and/or statins to respond anonymously, responses to the questionnaire(s) will be stored in their medical records. Data will then be extracted from the two systems [SystmOne and Egton Medical Information Systems (EMIS)] using unique system identifiers, that will be pseudonymised at the time of extraction. All patient pseudonymised information (including medical records system identifiers and responses to the questionnaire) will be extracted by the LTHT Researcher-Pharmacist following access provided by each participating General Practitioner (GP) Practice, based on searches built centrally by the Data Quality Team of the Leeds Clinical Commissioning Group (CCG).

Apart from the dissemination of findings based on the questionnaire, a training package for health professionals will be designed and delivered. The aim of the training is to combine and disseminate all findings of the project, raise awareness on real-world non-adherence prevalence and the common barriers to adherence, demonstrate the usefulness of routine adherence estimation and suggest tools to address non-adherence in daily practice. The objectives of this training will also consider the training needs of healthcare professionals locally, as per the healthcare professionals survey that has been designed and circulated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* having an active repeat prescription for a DOAC and/or a statin for at least 6 months prior to the date of data extraction
* a diagnosis of atrial fibrillation (AF) for those on a DOAC and of hypercholesterolemia for those on a statin (to justify the preventive nature of the treatments)

Exclusion Criteria:

* Patients with an active repeat prescription for a DOAC and/or a statin for less than 6 months prior to the date of data extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Charge from baseline adherence rates at 6 months | baseline, 6 months
  Barriers to DOAC and statin adherence that patients have chosen to disclose in the dedicated questionnaires. The rates of adherence based on repeat prescription data following the use of questionnaire(s) will also be compared with the individual rate before the use of questionnaire.
Frequency of reported adherence barriers | immediately after the intervention
  Commonly reported and less commonly reported barriers as a percentage of all responses

SECONDARY OUTCOMES:
Response rate, demographic and geographic variation | immediately after intervention
  Response rates in the integrated questionnaires within primary care systems

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouela Kampouraki, PhD, Study Chair — Leeds Teaching Hospitals Trust
Locations (1):
- Leeds Teaching Hospitals Trust, Leeds, West Yorkshire, United Kingdom